CLINICAL TRIAL: NCT04898179
Title: Targed Support for Patients Discharged After Hospitalization for SARS-CoV-2 Infection and Comorbidities. [ITALIAN. Supporto MIRATO ai Pazienti Dimessi Dopo un Ricovero Per Infezione da SARS-CoV-2 e comorbidità]
Brief Title: Support for COVID19 Patients at Home
Acronym: Mirato
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Auxologico Italiano (Other); Azienda Ospedaliera Bolognini di Seriate Bergamo (Other); Azienda Socio Sanitaria Territoriale di Bergamo (Unknown); University of Bergamo (Other)
Responsible Party: Sponsor
Other Study IDs: ICS Maugeri CE2455
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-09

CONDITIONS: COVID19 Patients
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telecare group: When discharged, patients will be followed at home by a telecare nursing and specialist teleconsultation program for 3 months. The key element of the program will be a structured nurse-managed telephone support and, when necessary, video consultations, to follow patients, for the first month. During these contacts, the nurse will conduct a standardized interview enquiring about the general clinical condition of the patient. In the case of any symptom or problem, the patient will be able to call the service. At the end of the third month, patients will contact again to check their clinical condition and to close the program. Patients will be provided with a pulse oximeter to measure O2 saturation.
  At the start and end of the program, patients were administered the SF-12 quality of life questionnaire.
  Interventions: Other: Telecare Group
- Control group: The patients in the control group will be followed by their general practitioner and they will be contacted after three months to check their clinical condition.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Telecare Group — Home-based telehealth program: telenursing and specialist teleconsultation
  Telemonitoring with a new pulse oximeter and specific App
  E-health platform
  Videoconference
  Groups: Telecare group
Other: Control group — Usual care
  Groups: Control group

SUMMARY:
The rapid spread and increase of acute respiratory infection cases caused by the novel SARS-CoV-2 coronavirus represent a major challenge for healthcare systems around the world. The shortage of facilities and medical personnel is a major problem in the face of a serious epidemic. The Lombardy Region, and in particular the territories of Milan, Bergamo and Brescia, was the most affected due to the rapid increase in cases and limited medical resources during the initial phase of the epidemic.

The collaboration between hospital and territory with integrated communication systems and the monitoring of patients with appropriate technological tools that include telemedicine, are fundamental to ensure the continuity of care and the sustainability of the health system, also significantly reducing the risk of contagion for health professionals.

DETAILED DESCRIPTION:
The MIRATO Project wants to test the remote health surveillance services and a telemonitoring program for patients discharged after a period of hospitalization for COVID19 caused by the new coronavirus SARS-CoV-2 and their comorbidities if present.

Patients discharged from hospitals still present in many cases breathing difficulties, bed rest symptoms and other disabilities related to the acute event. In addition, some patients are seeing rekindling of symptoms such as fever, dry cough, difficulty respiratory and blood desaturation into oxygen. These problems underline the need for procedures that allow us to safely discharge patients to be able to better follow their convalescence but also to be able to intervene quickly in the event of symptoms returning.

The purpose of the home health surveillance intervention will be:

* Monitor the evolution of the state of health with standardized tools based on scientific evidence
* Provide counselling support to help recovery
* Have certain and early identification of signs and symptoms related to a possible resumption of the COVID19 pathology and or to comorbidities
* Compare outcome results with case-control design three months after hospital discharge

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation for COVID19
* Patients discharged at home

Exclusion Criteria:

* Patient refusal
* Patients discharged at a nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized for COVID19
Sampling Method: Non-Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Re-hospitalisation at three months | 3 months
  Number of Re-hospitalisation registered at three months period in two groups
ER access at three months | 3 months
  Number of ER accesses registered at three months period in two groups
Death at three months | 3 months
  Number of death at three months in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Simonetta Scalvini, MD, Study Chair — Istituti Clinici Scientifici Maugeri
Locations (4):
- Italy (4):
  - Azienda Socio Sanitaria Territoriale (ASST) BERGAMO EST, Ospedale Bolognini di Seriate, Seriate, Bergamo
  - Ics Maugeri, Lumezzane, Brescia
  - Ics Maugeri, Tradate, Varese
  - Istituto Auxologico Italiano, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Word Health Organization. WHO Coronavirus Disease (COVID-19) Dashboard. Available at https://covid19.who.int 2020. (last accessed March 2021).
- [Background] Tebeje TH, Klein J. Applications of e-Health to Support Person-Centered Health Care at the Time of COVID-19 Pandemic. Telemed J E Health. 2021 Feb;27(2):150-158. doi: 10.1089/tmj.2020.0201. Epub 2020 Jul 31. PMID 32746750
- [Background] Doshi A, Platt Y, Dressen JR, Mathews BK, Siy JC. Keep Calm and Log On: Telemedicine for COVID-19 Pandemic Response. J Hosp Med. 2020 May;15(5):302-304. doi: 10.12788/jhm.3419. Epub 2020 Apr 1. No abstract available. PMID 32379036
- [Background] Tabacof L, Kellner C, Breyman E, Dewil S, Braren S, Nasr L, Tosto J, Cortes M, Putrino D. Remote Patient Monitoring for Home Management of Coronavirus Disease 2019 in New York: A Cross-Sectional Observational Study. Telemed J E Health. 2021 Jun;27(6):641-648. doi: 10.1089/tmj.2020.0339. Epub 2020 Oct 13. PMID 33232204
- [Background] Scalvini S, Bernocchi P, Zanelli E, Comini L, Vitacca M; Maugeri Centre for Telehealth and Telecare (MCTT). Maugeri Centre for Telehealth and Telecare: A real-life integrated experience in chronic patients. J Telemed Telecare. 2018 Aug;24(7):500-507. doi: 10.1177/1357633X17710827. Epub 2017 May 24. PMID 28537509
- [Background] Vitali A, Ghidotti A, Savoldelli A, Bonometti F, Rizzi C, Bernocchi P, Borghi G, Scalvini S. Definition of a Method for the Evaluation of Telemedicine Platforms in the Italian Context. Telemed J E Health. 2023 May;29(5):769-777. doi: 10.1089/tmj.2022.0326. Epub 2022 Oct 7. PMID 36206021
- [Result] Bernocchi P, Crotti G, Beato E, Bonometti F, Giudici V, Bertolaia P, Perger E, Remuzzi A, Bachetti T, La Rovere MT, Dalla Vecchia LA, Angeli F, Parati G, Borghi G, Vitacca M, Scalvini S. COVID-19 teleassistance and teleconsultation: a matched case-control study (MIRATO project, Lombardy, Italy). Front Cardiovasc Med. 2023 Aug 14;10:1062232. doi: 10.3389/fcvm.2023.1062232. eCollection 2023. PMID 37645519
- [Result] Bonometti F, Bernocchi P, Vitali A, Savoldelli A, Rizzi C, Scalvini S. Usability of a continuous oxygen saturation device for home telemonitoring. Digit Health. 2023 Aug 14;9:20552076231194547. doi: 10.1177/20552076231194547. eCollection 2023 Jan-Dec. PMID 37588158